CLINICAL TRIAL: NCT03821987
Title: Risk Stratification Directed Conditioning Regimen for Haploidentical HSCT in SAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Director of Institute Hematology,Peking University, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUIH-SAA
Record Dates: First submitted 2019-01-23; First posted 2019-01-30 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Aplastic Anemia; Stem Cell Transplant Complications; Engraft Failure
Keywords: haploidentical transplantation; aplastic anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — fludarabine; Busulfan; Cyclophosphamide; thymoglobulin

STUDY DESIGN:
Intervention Model Description: Patients enrolled in this study would receive Bu (IV)0.8mg/kg Q6hx2d,Fludarabine 30mg/m2x5d ,CTX(cyclophosphamide) 25mg/kg/dx4d,rATG (thymoglobulin,Sang Stat,France) 2.5mg/kg/dx4d.
  BM or Blood samples from patients were obtained to assess engraftment and chimerism after HSCT. The time point that we monitored BM or blood samples included at 1 month,2 months, 3 months,6 months, 9 months and 1year,2years,3years 5 years after HSCT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BFCA regimen (Experimental): Detail: Patients enrolled in this study would receive Busulfan(B) (IV)0.8mg/kg Q6hx2d,Fludarabine(F) 30mg/m2x5d ,cyclophosphamide(C) 25mg/kg/dx4d,thymoglobulin (A :rATG ,Sang Stat,France) 2.5mg/kg/dx4d.
  BM or Blood samples from patients were obtained to assess engraftment and chimerism after HSCT. The time point that we monitored BM or blood samples included at 1 month,2 months, 3 months,6 months, 9 months and 1year,2years,3years 5 years after HSCT.
  Interventions: Drug: Fludarabine

INTERVENTIONS:
Drug: Fludarabine — Patients enrolled in this study would receive Bu (IV)0.8mg/kg Q6hx2d,Fludarabine 30mg/m2x5d ,CTX (cyclophosphamide) 25mg/kg/dx4d,rATG (thymoglobulin,Sang Stat,France) 2.5mg/kg/dx4d.
  Other Names: Busulfan; Cyclophosphamide; Thymoglobulin

SUMMARY:
The haplotype HSCT system including Bu(0.8mg/kg Q6hx2d)CTX(50mg/kgx4d)rATG(2.5mg/kgx4d) , established in Institute of Hematology of Peking University ,has been evaluated to be effective for acquired SAA.But some patients with high risk factors may not tolerate CTX 200mg/kg,alternative conditioning regimen including Bu/Fludarabine/dercreased CTX was studied in this trial.

DETAILED DESCRIPTION:
Patients enrolled in this study would receive Bu (IV)0.8mg/kg Q6hx2d,Fludarabine 30mg/m2x5d ,CTX(cyclophosphamide) 25mg/kg/dx4d,rATG (thymoglobulin,Sang Stat,France) 2.5mg/kg/dx4d.

BM or Blood samples from patients were obtained to assess engraftment and chimerism after HSCT. The time point that investigators monitor BM or blood samples at 1 month,2 months, 3 months,6 months, 9 months and 1year,2years,3years 5 years after HSCT.

ELIGIBILITY:
A：inclusion criteria

1. Patients diagnosed as acquired severe aplastic anemia(SAA) /very vSAA
2. patients with age 3-55 years
3. patients have no matched sibling donor
4. Patients have no matched unrelated donor
5. patients have no severe infection
6. Patients have no severe organ dysfunction
7. patients have risk factors of potential intolerance to previous condition regimen including BuCy(200mg/kg)and ATG
8. Consent form signed

B. Exclusion criteria ：

1. patients with congenital SAA/vSAA
2. patients with age< 3years or >55 years
3. patients with matched sibling donor
4. patients with matched URD
5. patients with severe infection
6. patients with severe organ dysfunction
7. pregnancy women
8. no Consent form signed

Ages: 3 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
1 year cumulative incidence overall survival | 1 year post HSCT
  Tne cumulative incidence of overall survival at 1 year post HSCT

SECONDARY OUTCOMES:
one month Transplantation related mortality | 1 month post HSCT
  Tne cumulative incidence of transplantation related motality at 1 month post HSCT
Engraftment | 1 month post HSCT
  Tne cumulative incidence of engraftment at 1 moths post HSCT
0ne month regimen-related toxicity | 1 month post HSCT
  Tne cumulative incidence of regimen related toxicity at 1 month post HSCT
aGVHD | 100 days post HSCT
  Tne cumulative incidence of acute GVHD at Day 100 post HSCT
failure-free survival | 1 year post HSCT
  The cumulative incidence of failure-free survival at 1year post HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, Prof., Principal Investigator — Peking Universiy Institute of Hematology,People's Hospital Pekiking Universiyy
Locations (1):
- Peking University Institute of Hematology,People's hospital Peking University, Beijing, Beijing Municipality, China